CLINICAL TRIAL: NCT02569541
Title: An Open-Label, Non-Randomized, Single-Arm, Multi-Center Study to Evaluate Oral Sodium Fusidate (CEM-102) for the Treatment of Staphylococcal Bone or Joint Infections in Subjects for Whom Chronic Antibiotic Suppressive Therapy is Indicated
Brief Title: Oral Sodium Fusidate (CEM-102) for the Treatment of Staphylococcal Bone or Joint Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Arrevus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE06-302
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Refractory Bone or Joint Infections
Keywords: fusidic acid; prosthetic joint infections; bone infections; osteomyelitis
MeSH Terms: conditions — Osteomyelitis | interventions — Fusidic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CEM-102 (Sodium fusidate) (Experimental): 1500 mg by mouth every 12 hours for 2 doses, then 600 mg by mouth every 12 hours thereafter, until end of therapy:
  * 6 months of treatment; or
  * 24 months of treatment (if continued on chronic suppressive therapy)
  Interventions: Drug: sodium fusidate

INTERVENTIONS:
Drug: sodium fusidate
  Other Names: CEM-102; fusidic acid

SUMMARY:
To evaluate the safety and effectiveness of oral sodium fusidate (CEM-102) as chronic antibiotic for the treatment of bone or joint infections.

DETAILED DESCRIPTION:
Prospective, open-label, non-randomized, single-arm trial to evaluate the safety and effectiveness of CEM-102 for chronic antibiotic suppressive therapy of bone or joint infections. Subjects enrolling in this study must have a refractory staphylococcal bone or joint infection that requires suppressive antibiotic therapy (e.g. having an infection that cannot be managed by complete removal of the infected bone or foreign material, a refractory infection not responding to previous treatment, or not being a candidate for long-term intravenous antibiotic therapy).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 12 and 18 years must weigh >60 kg
* Bone or joint infection due to an inclusionary pathogen demonstrated from a culture from samples obtained within 6 weeks prior to enrollment
* Not a candidate, as determined by the Investigator, for suitable alternative therapy
* After completion of 1-2 weeks of the companion antibiotic, must be a suitable candidate for CEM-102 monotherapy for chronic treatment

Exclusion Criteria:

* Requires concomitant treatment with OATP1B1 and OATP1B3 substrates, in particular, statins (HMG-CoA reductase inhibitors)
* Known severe renal impairment, as indicated by estimated CrCl <30 mL/min (by Cockcroft-Gault calculation)
* Evidence of significant liver disease: ALT >3 × ULN or direct bilirubin >ULN; known cirrhosis with decompensation (i.e. Child-Pugh Class B or C disease)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2017-10-17 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dobbins, MD, PhD, Study Director — Melinta Therapeutics, Inc.
Locations (19):
- United States (19):
  - Fountain Valley, California
  - San Dimas, California
  - Sylmar, California
  - Torrance, California
  - Tamarac, Florida
  - Springfield, Illinois
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Butte, Montana
  - Somers Point, New Jersey
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Haverford, Pennsylvania
  - Malvern, Pennsylvania
  - Philadelphia, Pennsylvania
  - Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CEM-102 (Sodium Fusidate): 1500 mg by mouth every 12 hours for 2 doses, then 600 mg by mouth every 12 hours thereafter, until end of therapy:
  * 6 months of treatment; or
  * 24 months of treatment (if continued on chronic suppressive therapy)
  sodium fusidate
Period: Overall Study
Arm/Group | CEM-102 (Sodium Fusidate)
Started | 30
Completed | 9
Not Completed | 21

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all subjects who provided informed consent, met all eligibility criteria, and were enrolled in the study.
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Height [Mean (Standard Deviation); unit: cm] | 174.5 (11.54)
Weight [Mean (Standard Deviation); unit: kg] | 87.4 (22.12)
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.7 (6.79)
Infection Type and Location [Count of Participants; unit: Participants]
  Osteomyelitis | 4
  Chronic septic arthritis - knee | 1
  Prosthetic joint infection - knee | 11
  Prosthetic joint infection - hip | 4
  Prosthetic joint infection - shoulder | 1
  Prosthetic joint infection - other | 4
  Other orthopedic hardware | 5
Risk Factors for BJI [Count of Participants; unit: Participants]
  Rheumatoid Arthritis | 3
  Diabetes Mellitis | 8
  Decubitis ulcers from Immobility | 4
  Previous PJI in Another Anatomical Location | 4
Baseline Pathogen [Count of Participants; unit: Participants]
  Staphylococcus aureus (MSSA) | 12
  Staphylococcus aureus (MRSA) | 10
  Staphylococcus epidermidis | 4
  coagulase-negative Staphylococcus | 3
  Corynebacterium striatum/simulans | 2
  Cutibacterium acnes | 1
  Streptococcus agalactiae | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success at 6 Months
Description: Number of participants in the intent to treat (ITT) analysis set who meet all the criteria for clinical success at the 6-Month Visit.
  Clinical success was defined to occur when subjects met all of the following criteria: 1) Subject was not hospitalized due to worsening of the study-qualifying orthopedic infection. 2) Subject did not undergo a definitive surgical procedure (such as amputation). 2) No additional antibiotics (after completion of companion antibiotics) are required for treatment of the orthopedic infection due to the inclusionary pathogen. 3) Wound is closed, or the open area decreased in size (L x W) and, if a skin graft was done, the graft remains viable without evidence of infection. 4) No purulent discharge from the surgical wound, or new or recurring sinus tract. 5) No worsening of redness, tenderness, or swelling at the primary infection site. 5) No bacteremia
Time Frame: 6 months after start of treatment
Population: ITT Population - all subjects who provided informed consent, met all eligibility criteria, and were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Participants
  Clinical Success | 18
  Clinical Failure | 9
  Indeterminate | 3

2. Secondary Outcome: Safety and Tolerability
Description: Number of participants with TEAEs, SAEs, deaths, and discontinuations due to AEs.
  Treatment-emergent adverse events, defined as events with a start date on or after the initiation of study drug through 28 days after the last dose of study drug, are reported.
Time Frame: Entire study period - up to 24 months
Population: Safety population - all enrolled subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Participants
  Treatment Emergent AE (TEAE) | 29
  Severe TEAE | 12
  TEAE Related to Study Drug | 7
  TEAE Leading to Study Discontinuation | 9
  TEAE Leading to Study Drug Discontinuation | 12
  TE Serious Adverse Event (SAE) | 15
  TE SAE with outcome of death | 0
  TE SAE Related to Study Drug | 0
  TE SAE Leading to Study Discontinuation | 7
  TE SAE Leading to Study Drug Discontinuation | 9

3. Secondary Outcome: Clinical Success at 9 Months
Description: Number of participants in the ITT analysis set who meet all the criteria for clinical success at the 9-Month Visit.
  Clinical success was defined to occur when subjects met all of the following criteria: 1) Subject was not hospitalized due to worsening of the study-qualifying orthopedic infection. 2) Subject did not undergo a definitive surgical procedure (such as amputation). 2) No additional antibiotics (after completion of companion antibiotics) are required for treatment of the orthopedic infection due to the inclusionary pathogen. 3) Wound is closed, or the open area decreased in size (L x W) and, if a skin graft was done, the graft remains viable without evidence of infection. 4) No purulent discharge from the surgical wound, or new or recurring sinus tract. 5) No worsening of redness, tenderness, or swelling at the primary infection site. 5) No bacteremia
Time Frame: 9 months after start of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Participants
  Clinical Success | 15
  Clinical Failure | 11
  Indeterminate | 4

4. Secondary Outcome: Clinical Success at 12 Months
Description: Number of participants in the ITT analysis set who meet all the criteria for clinical success at the 12-Month Visit.
  Clinical success was defined to occur when subjects met all of the following criteria: 1) Subject was not hospitalized due to worsening of the study-qualifying orthopedic infection. 2) Subject did not undergo a definitive surgical procedure (such as amputation). 2) No additional antibiotics (after completion of companion antibiotics) are required for treatment of the orthopedic infection due to the inclusionary pathogen. 3) Wound is closed, or the open area decreased in size (L x W) and, if a skin graft was done, the graft remains viable without evidence of infection. 4) No purulent discharge from the surgical wound, or new or recurring sinus tract. 5) No worsening of redness, tenderness, or swelling at the primary infection site. 5) No bacteremia
Time Frame: 12 months after start of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Participants
  Clinical Success | 10
  Clinical Failure | 15
  Indeterminate | 5

5. Secondary Outcome: Clinical Success at 15 Months
Description: Number of participants in the ITT analysis set who meet all the criteria for clinical success at the 15-Month Visit.
  Clinical success was defined to occur when subjects met all of the following criteria: 1) Subject was not hospitalized due to worsening of the study-qualifying orthopedic infection. 2) Subject did not undergo a definitive surgical procedure (such as amputation). 2) No additional antibiotics (after completion of companion antibiotics) are required for treatment of the orthopedic infection due to the inclusionary pathogen. 3) Wound is closed, or the open area decreased in size (L x W) and, if a skin graft was done, the graft remains viable without evidence of infection. 4) No purulent discharge from the surgical wound, or new or recurring sinus tract. 5) No worsening of redness, tenderness, or swelling at the primary infection site. 5) No bacteremia
Time Frame: 15 months after start of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Participants
  Clinical Success | 8
  Clinical Failure | 17
  Indeterminate | 5

6. Secondary Outcome: Clinical Success at 18 Months
Description: Number of participants in the ITT analysis set who meet all the criteria for clinical success at the 18-Month Visit.
  Clinical success was defined to occur when subjects met all of the following criteria: 1) Subject was not hospitalized due to worsening of the study-qualifying orthopedic infection. 2) Subject did not undergo a definitive surgical procedure (such as amputation). 2) No additional antibiotics (after completion of companion antibiotics) are required for treatment of the orthopedic infection due to the inclusionary pathogen. 3) Wound is closed, or the open area decreased in size (L x W) and, if a skin graft was done, the graft remains viable without evidence of infection. 4) No purulent discharge from the surgical wound, or new or recurring sinus tract. 5) No worsening of redness, tenderness, or swelling at the primary infection site. 5) No bacteremia
Time Frame: 18 months after start of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Participants
  Clinical Success | 8
  Clinical Failure | 16
  Indeterminate | 6

7. Secondary Outcome: Clinical Success at 21 Months
Description: Number of participants in the ITT analysis set who meet all the criteria for clinical success at the 21-Month Visit.
  Clinical success was defined to occur when subjects met all of the following criteria: 1) Subject was not hospitalized due to worsening of the study-qualifying orthopedic infection. 2) Subject did not undergo a definitive surgical procedure (such as amputation). 2) No additional antibiotics (after completion of companion antibiotics) are required for treatment of the orthopedic infection due to the inclusionary pathogen. 3) Wound is closed, or the open area decreased in size (L x W) and, if a skin graft was done, the graft remains viable without evidence of infection. 4) No purulent discharge from the surgical wound, or new or recurring sinus tract. 5) No worsening of redness, tenderness, or swelling at the primary infection site. 5) No bacteremia
Time Frame: 21 months after start of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Participants
  Clinical Success | 6
  Clinical Failure | 17
  Indeterminate | 7

8. Secondary Outcome: Clinical Success at 24 Months
Description: Number of participants in the ITT analysis set who meet all the criteria for clinical success at the 24-Month Visit.
  Clinical success was defined to occur when subjects met all of the following criteria: 1) Subject was not hospitalized due to worsening of the study-qualifying orthopedic infection. 2) Subject did not undergo a definitive surgical procedure (such as amputation). 2) No additional antibiotics (after completion of companion antibiotics) are required for treatment of the orthopedic infection due to the inclusionary pathogen. 3) Wound is closed, or the open area decreased in size (L x W) and, if a skin graft was done, the graft remains viable without evidence of infection. 4) No purulent discharge from the surgical wound, or new or recurring sinus tract. 5) No worsening of redness, tenderness, or swelling at the primary infection site. 5) No bacteremia
Time Frame: 24 months after start of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CEM-102 (Sodium Fusidate)
Number analyzed (Participants) | 30
Participants
  Clinical Success | 7
  Clinical Failure | 17
  Indeterminate | 6

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events are reported for members of the Safety Population, comprised of enrolled subjects who received at least 1 dose of study drug. Treatment-emergent adverse events, defined as events with a start date on or after the initiation of study drug through 28 days after the last dose of study drug, are reported.
Arm/Group | CEM-102 (Sodium Fusidate)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 15/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEM-102 (Sodium Fusidate) (N=30)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 4 (4)
Diverticulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Yellow nail syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Abscess drainage (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEM-102 (Sodium Fusidate) (N=30)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Vision blurred (Eye disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 4 (4)
Peripheral swelling (General disorders) | 4 (4)
Pyrexia (General disorders) | 4 (4)
Cellulitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 9 (9)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2)
International normalised ratio increased (Investigations) | 2 (2)
Weight decreased (Investigations) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the right to first publication of results, which would be made in conjunction with the PIs from all appropriate sites. Thereafter, PIs may publish results provided the PI submits the proposed publication to the Sponsor for review at least 60 days prior to the date of the proposed publication. The Sponsor may remove information that is considered confidential and/or proprietary and delay the proposed publication for an additional 60 days to enable filing of patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT02569541/Prot_SAP_000.pdf